CLINICAL TRIAL: NCT02030522
Title: Prospective Cohort Study of Accelerated Resolution Therapy (ART) for Treatment of Military Psychological Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013717
Record Dates: First submitted 2013-11-04; First posted 2014-01-08 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2014-12

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: Post-traumatic stress disorder; PTSD; Accelerated Resolution Therapy; Military; Veterans; Exposure therapy; Eye movements
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective Treatment Cohort of ART (Experimental): The target population (n=200) of persons treated with the intervention, Accelerated Resolution Therapy, will consist of U.S. service members and veterans who have symptoms indicative of a current diagnosis of PTSD. No age limit or duration of symptoms of PTSD will be imposed for study eligibility, and it is anticipated that most, if not all, of eligible and enrolled participants will have had prior deployments to conflicts dating back to the 1970s, including the Vietnam War, Persian Gulf conflict, and wars in Iraq and Afghanistan. No person will be excluded on the basis of race, ethnicity, gender, or disability.
  Interventions: Behavioral: Accelerated Resolution Therapy (ART)

INTERVENTIONS:
Behavioral: Accelerated Resolution Therapy (ART) — The ART protocol will be delivered in 2-5 sessions. Imaginal Exposure (IE) will be used whereby service members and veterans will be asked to recall (verbally or non-verbally) details of the traumatic event(s) while focusing their attention on physiological sensations, thoughts, and emotions. This short period of exposure to the memory will be followed by identification and diminishment of the emergence of any uncomfortable emotional or somatic symptoms. Imagery Rescripting (IR) will be used to change (replace) negative traumatic images to positive images. The service member/veteran will imagine and play out an affectively-driven solution to change sensory components of the memory, as if they were the "director of the movie" of the memory they are working on.

SUMMARY:
This is a prospective cohort treatment intervention study (n=200) whereby U.S. service members and veterans with symptoms of PTSD will undergo 2-5 sessions of ART delivered by Florida licensed mental health professionals trained in ART. The 3 study aims are to: (i) evaluate among U.S. service members and veterans overall, and within specific subgroups, the magnitude of change in symptoms of PTSD following treatment with ART; (ii) evaluate the sustainability of treatment response with ART; and (iii) evaluate the cost effectiveness of ART compared to prolonged exposure (PE) therapy in the treatment of symptoms of PTSD.

DETAILED DESCRIPTION:
This study entitled "Prospective Cohort Study of Accelerated Resolution Therapy (ART) for Treatment of Military Psychological Trauma" is a prospective cohort treatment intervention study (n=200) whereby U.S. service members and veterans with symptoms of PTSD will undergo 2-5 sessions of ART delivered by Florida licensed mental health professionals trained in ART. Clinical assessments will be conducted pre-treatment, post-treatment (approximately 2 weeks after study entry), and at 6-month follow-up (self-report questionnaires). The study aligns with the USF College of Nursing POWER initiative by seeking to expand the science base of effective treatment of service members and veterans with impaired psychological status. The study rationale is to: (i) demonstrate that ART is a brief, effective, and safe treatment for military-related PTSD including military sexual trauma (MST) and among service members with PTSD refractory to previous psychotherapy; (ii) provide evidence of the sustainability of clinical response 6-months after treatment completion; (iii) provide evidence that ART is a cost effective treatment for PTSD compared to current therapies formally endorsed by the VA and DoD; and (iv) develop the infrastructure for expansion of the ART protocol and science base, including national and international treatment settings, expanded patient populations, expanded clinical services, and mechanistic studies of ART. The target population (n=200) will consist of U.S. service members and veterans who have symptoms indicative of a current diagnosis of PTSD. Oversampling will occur for participants with a history of MST (minimum n=60) and/or PTSD refractory to prior psychotherapy (minimum n=60). No age limit or duration of symptoms of PTSD will be imposed for study eligibility, and it is anticipated that most, if not all, of eligible and enrolled participants will have had prior deployments to conflicts dating back to the 1970s, including the Vietnam War, Persian Gulf War, and the more recent wars in Iraq and Afghanistan. Demographic and medical history data will be collected along with details of prior military service including service branch, deployment location(s) and type of trauma(s). Participants will complete the 7-item Combat Exposure Scale and 3-item Brief Traumatic Brain Injury Screen. To evaluate treatment response, measures completed at entry, post-treatment, and 6 months will include: 17-item PCL-M (PTSD Checklist), 125-item Psychiatric Diagnostic Screening Questionnaire, 18-item Brief Symptom Inventory (BSI), 34-item Clinical Outcomes in Routine Evaluation (CORE-OM) scale, Medical Outcome Study Short Form-36, 20-item Center for Epidemiological Studies Depression Scale (CES-D), 21-item State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA), 22-item Trauma-Related Guilt Inventory (TRGI), and use of medications. The study will be conducted over a 24-month period.

ELIGIBILITY:
Inclusion Criteria:

* U.S. service member or veteran with prior deployment(s) to a major conflict zone(s)(e.g. Vietnam War, Persian Gulf conflict, and wars in Iraq and Afghanistan).
* Symptoms indicative of current PTSD. This includes: (i) score of >40 on the PCL-M Checklist; (ii) endorsement of PCL-M symptoms rated as "Moderately" or above as follows: at least 1 B item (questions 1-5), 3 C items (questions 6-12), and at least 2 D items (questions 13-17); and (iii) scoring positive on the PTSD subscale of the Psychiatric Diagnostic Screening Questionnaire.
* Ability to read and speak English to complete survey questions.
* Denial of suicidal ideation or intent, including homicidal ideation or intent, and no evidence of psychotic behavior or being in psychological crisis.

Exclusion Criteria:

* Brain injury prohibiting speech, writing, and purposeful actions.
* Currently engaged in another PTSD psychotherapy treatment intervention. Screening therapist will determine eligibility based on the type of psychotherapy and medications the participant is receiving.
* Major psychiatric disorder (e.g. bipolar disorder) concomitant to symptoms of psychological trauma and deemed likely to interfere with treatment delivery.
* Currently undergoing substance abuse treatment (alcohol and/or drug).
* Any medical condition that, in the judgment of the Principal Investigator and/or ART clinician, may place the individual at high risk due to a potential heightened emotional reaction (e.g. previous heart attack, seizure disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
17-item PTSD Checklist-Military (PCL-M) | Change from pre-treatment to post-treatment and 6-month follow-up
  The PCL-M Checklist is a self-administered 17-item scale that corresponds to key symptoms of PTSD. Reliability estimates range from .92 to .97, and the PCL has been validated in both civilians and veterans. Respondents rate how much they were "bothered by that problem in the past month". Items are rated on a 5-point scale ranging from 1 ("not at all") to 5 ("extremely"). The PCL can be scored in several different ways. A total score (range 17-85) can be obtained by summing the scores from each of the 17 items. Cutoff scores for a probable PTSD diagnosis have been validated for some populations, but may not generalize to other populations. A second way to score the PCL is to follow the DSM-IV criteria. Strong convergent validity has been reported.

SECONDARY OUTCOMES:
Brief Symptom Inventory | Change from pre-treatment to post-treatment and 6-month follow-up
  The 18-item Brief Symptom Inventory (BSI) is a shortened version of the Symptom Checklist 90-Revised (SCL-R-90) designed to measure clinically relevant psychological symptoms in adolescents and adults. This instrument encompasses 3 factors: Somatization, Depression, and Anxiety, along with a Global Severity Index. This inventory shows satisfactory reliability indexes, both for the individual factors (ranging from 0.74 to 0.84) and the Global Severity Index (0.89).
Center for Epidemiological Studies Depression Scale | Change from pre-treatment to post-treatment and 6-month follow-up
  The 20-item Centers for Epidemiological Studies Depression Scale (CES-D) is a widely used self-report scale that measures current level of depressive symptomatology with an emphasis on depressed mood during the past week. The CES-D incorporates the main symptoms of depression and was derived from five validated depression scales including the Beck Depression Inventory (BDI). It is freely available in the public domain, has been validated in community and primary care populations, and has good test-retest reliability (range 0.84 to 0.92).
Clinical Outcomes in Routine Evaluation | Change from pre-treatment to post-treatment and 6-month follow-up
  The 34-item Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) is a generic measure of psychological distress, which is pan-theoretical (i.e., not associated with a school of therapy), pan-diagnostic (i.e. not focused on a single presenting problem), and draws upon the views of what practitioners consider to be the most important generic aspects of psychological well-being health to measure. The CORE-OM comprises 4 domains: well-being (4 items), symptoms (12 items), functioning (12 items), and risk (6 items). Internal consistency coefficients range from 0.70 to 0.97 across all domains and among primary and secondary care settings.
Medical Outcome Study Short Form-36 (SF-36) | Change from pre-treatment to post-treatment and 6-month follow-up
  The Medical Outcome Study Short Form-36 (SF-36) is an established, widely used measure for constructing a health utility index. It is a self-report 36-item health status measure that uses a Likert-type response format. The eight subscales of SF-36 include the domains of role limitations with regard to physical health, emotional health, energy/fatigue, emotional well-being, social functioning, pain, and general health, along with a general scale on physical functioning. Subscale scores range from 0 to 100 with higher scores indicating a more favorable health status. Estimates of internal consistency reliability range from 0.62 to 0.94; the majority of scores have exceeded 0.80. Test-retest reliability estimates range from 0.43 to 0.90. Factor analysis indicates two dimensions of the instrument, physical and mental health status, that account for 82% of the reliable variance of the measure.
State-Trait Inventory for Cognitive and Somatic Anxiety | Change from pre-treatment to post-treatment and 6-month follow-up
  The 21-item State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) is designed to assess cognitive and somatic symptoms of anxiety as they pertain to one's mood in the moment (state) and in general (trait). It takes an estimated 6 minutes to complete. The STICSA is a reliable and valid measure of state and trait cognitive and somatic anxiety, with coefficients ranging from 0.87 to 0.90.
Pittsburgh Sleep Quality Index | Change from pre-treatment to post-treatment and 6-month follow-up
  The 15-item Pittsburgh Sleep Quality Index (PSQI) measures quality and patterns of sleep in adults. It takes an estimated 3 to 6 minutes to complete. A global PSQI score greater than 5 has yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% (kappa = 0.75, p<0.001) in distinguishing good and poor sleepers. Internal consistency reliability has been estimated to range from .77 to .81.
Trauma-Related Guilt Inventory | Change from pre-treatment to post-treatment and 6-month follow-up
  The 22-item Trauma Related Guilt Inventory (TRGI) assesses event-focused, trauma-related guilt. The inventory has high internal consistency and adequate temporal stability, and its scales and subscales significantly correlate with measures of guilt and PTSD, depression, and adjustment. Reliability coefficients range from 0.73 to 0.91. The time to complete the inventory is estimated to be 6 minutes.
Pain Outcomes Questionnaire | Change from pre-treatment to post-treatment and 6-month follow-up
  The 20-item Pain Outcomes Questionnaire (POQ) - Short Form is a reliable and valid instrument that contains 19 primary pain items that are rated on an 11-point (0-10) Likert-type scale and one demographic question. In addition to a total pain score, six subscale scores can be calculated that correspond to: pain intensity (1 item), pain-related impairment in mobility (4 items), pain-related impairment in performing activities of daily living (4 items), sense of impairment in activity and energy levels (3 items), dysphoric affect and associated symptoms (5 items), and pain-related fear and avoidance (2 items).
Psychiatric Diagnostic Screening Questionnaire | Change from pre-treatment to post-treatment and 6-month follow-up
  The 125-item Psychiatric Diagnostic Screening Questionnaire (PDSQ) is used to screen for Axis I disorders and global assessment of psychopathology. This instrument has been validated against diagnostic criteria and interview-derived diagnoses over the course of 10 years and more than 3,000 administrations. It can be quickly hand scored to obtain a total score (which functions as a global indicator of psychopathology) plus subscale scores for 13 disorders: major depressive disorder (MDD), generalized anxiety disorder, panic disorder, PTSD, alcohol abuse/dependence, drug abuse/dependence, psychosis, bulimia/binge-eating disorder, somatization disorder, obsessive-compulsive disorder, social phobia, hypochondriasis, and agoraphobia.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Kip, Ph.D., Principal Investigator — University of South Florida
Locations (8):
- United States (8):
  - Homeless Emergency Project (HEP), Clearwater, Florida
  - Veterans Alternative Therapy Center, Holiday, Florida
  - Life Renewal Counseling, Jupiter, Florida
  - Pasco County Detention Center, Land O' Lakes, Florida
  - Supportive Services for Veterans Families, New Port Richey, Florida
  - Gilstrap & Associates, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Cornerstone Counseling, Auburn, Maine

REFERENCES:
- [Background] Kip KE, Sullivan KL, Lengacher CA, Rosenzweig L, Hernandez DF, Kadel R, Kozel FA, Shuman A, Girling SA, Hardwick MJ, Diamond DM. Brief treatment of co-occurring post-traumatic stress and depressive symptoms by use of accelerated resolution therapy((R)). Front Psychiatry. 2013 Mar 8;4:11. doi: 10.3389/fpsyt.2013.00011. eCollection 2013. PMID 23482431
- [Background] Kip KE, Rosenzweig L, Hernandez DF, Shuman A, Diamond DM, Girling SA, Sullivan KL, Wittenberg T, Witt AM, Lengacher CA, Anderson B, McMillan SC. Accelerated Resolution Therapy for treatment of pain secondary to symptoms of combat-related posttraumatic stress disorder. Eur J Psychotraumatol. 2014 May 7;5. doi: 10.3402/ejpt.v5.24066. eCollection 2014. PMID 24959325
- [Background] Kip KE, Shuman A, Hernandez DF, Diamond DM, Rosenzweig L. Case report and theoretical description of accelerated resolution therapy (ART) for military-related post-traumatic stress disorder. Mil Med. 2014 Jan;179(1):31-7. doi: 10.7205/MILMED-D-13-00229. PMID 24402982
- [Background] Kip KE, Rosenzweig L, Hernandez DF, Shuman A, Sullivan KL, Long CJ, Taylor J, McGhee S, Girling SA, Wittenberg T, Sahebzamani FM, Lengacher CA, Kadel R, Diamond DM. Randomized controlled trial of accelerated resolution therapy (ART) for symptoms of combat-related post-traumatic stress disorder (PTSD). Mil Med. 2013 Dec;178(12):1298-309. doi: 10.7205/MILMED-D-13-00298. PMID 24306011
- See also: Huffington Post Commentary on Accelerated Resolution Therapy — http://m.huffpost.com/us/entry/4093413